CLINICAL TRIAL: NCT06310226
Title: Characterizing Functional MRI Phenotypes in Response to Spinal Cord Stimulation in Chronic Low Back Pain
Brief Title: Phenotyping Response to Spinal Cord Stimulation in Chronic Low Back Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Daniel Lu, MD, PhD, Principal Investigator, Neuroplasticity and Repair Laboratory, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 23-000347
Record Dates: First submitted 2024-03-04; First posted 2024-03-15 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-06

CONDITIONS: Chronic Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Responders to spinal cord stimulation (Experimental): Patients with chronic low back pain, with >50% pain reduction in response to spinal cord stimulation
  Interventions: Device: Epidural electrical spinal cord stimulator
- Non-responders to spinal cord stimulation (Experimental): Patients with chronic low back pain, with minimal to no pain reduction in response to spinal cord stimulation
  Interventions: Device: Epidural electrical spinal cord stimulator

INTERVENTIONS:
Device: Epidural electrical spinal cord stimulator — Epidural electrical spinal cord stimulator turned on vs. turned off

SUMMARY:
Chronic low back pain (CLBP) is a debilitating condition and costly to treat. Long-term drug treatment often fails due to habituation, breakthrough of pain, or adverse effects of drug treatment. Opioid use to manage this pain has contributed to the opioid epidemic. Spinal cord stimulators have emerged as a promising treatment and reduces reliance on drugs. However, response to spinal cord stimulation (SCS) is unpredictable. It is difficult to predict which patients will respond positively to SCS because the physiological mechanism for treatment responsiveness is unclear. Therefore, the aim of this study is to investigate how spinal cord stimulators affect functional measures in patients with CLBP, including functional MRI, neurophysiology, gait analysis, and questionnaires. The results of this study can lead to the widespread adoption of spinal cord stimulators as a safe and effective therapy for CLBP, reducing the reliance on opioids and mitigating the opioid epidemic's impact.

DETAILED DESCRIPTION:
Electrical stimulation of neural tissues can be effective and reduce reliance on drugs, and epidural spinal cord stimulation (SCS) is often used to treat chronic low back pain (CLBP). Despite a half-century of clinical use, the mechanism of action of SCS remains unclear. Many patients fail to respond to SCS, and lacking a thorough understanding of the biological processes underlying SCS, there are no established predictors of treatment response to SCS. The application of SCS today is dependent on an empirical trial-and-error approach, which is expensive, time consuming, and frustrating for the patient. Even with the advent of improved stimulation technology and novel stimulation strategies (e.g., high frequency, burst stimulation, etc.), device failure rates remain high. CLBP is a multi-faceted process involving abnormal processing in the sensorimotor cortices, prefrontal cortex, insula, thalamus, limbic system, cerebellum, and brainstem nuclei including the periaqueductal gray, locus coeruleus, and dorsal raphe nuclei, all of which function in the context of myriad individual psychosocial factors.

The goal of this study is to develop a quantitative description of the neurophysiological processes associated with the sensation of pain and identify the signature(s) of pain, the neurophysiological pain connectome (NPC), that may guide treatment more effectively. The investigators hypothesize CLBP is marked by a pattern of pathological activity resulting from interactions among different brain networks. The investigators theorize the spatiotemporal patterns of activity among these networks, which are reflected in the NPC, are maladaptive and expressed as abnormal cognitive, affective, and sensorimotor expressions of chronic pain. Because CLBP is a complex disorder, a fundamentally different approach is necessary to assess the many facets of the NPC using comprehensive multi-modal assessments.

Investigators will use: 1. functional and diffusion MRI to quantify brain functional and microstructural connectivity; 2. electroencephalography (EEG); 3. gait kinematics; and 4. electrophysiology (somatosensory evoked potential, SSEP and pain-related evoked potentials, PREPs) to evaluate the neurotransmission of pain. Investigators will then correlate patterns in the NPC with a range of patient-reported outcomes including the domains of the PROMIS questionnaires, and combine this information to generate models based on the patterns in the NPC most closely associated with specific aspects of pain and the patient experience.

ELIGIBILITY:
Inclusion Criteria:

* Able to give informed consent for participation in the trial and be able to comply with study-related requirements, procedures, and visits
* Male or female, between the ages of 18 and 80 years (inclusive)
* Current self-report of chronic low back pain (pain between the lower posterior margin of the rib cage and the horizontal gluteal fold), which has persisted for > the past 3 months AND has resulted in pain on > 50% of days in the past 6 months* (*Chronic low back pain criteria as defined by the NIH Pain Consortium Research Task Force (RTF) and BACPAC Minimum Dataset Working Group)
* Already undergoing spinal cord stimulator treatment for chronic low back pain
* Able to use their lower extremities
* Able to tolerate fMRI and neurophysiological evaluation

Exclusion Criteria:

* Significant decision-making incapacity preventing informed consent
* Any medical condition that could interfere with study procedures, accurate pain reporting, and/or confound evaluation of study endpoints, as determined by the Investigator.
* Lifetime history of psychiatric disorder (schizophrenia, bipolar disorder with psychotic features, or other psychotic disorder), or current suicidal ideation
* Any stimulation device and/or implant other than a spinal cord stimulator, such as a drug pump, pacemaker, deep brain stimulator (DBS), or sacral nerve stimulator (SNS)
* Life expectancy of less than 1 year
* Pregnant or nursing (if female and sexually active, patient must be using a reliable form of birth control, be surgically sterile, or be at least 2 years post-menopausal)
* Any documented history of substance abuse (narcotics, alcohol, etc.) or substance dependency (not including marijuana use)
* Participation in another clinical trial currently or within the past 30 days
* Current treatment with electroconvulsive therapy (ECT) or transcranial magnetic stimulation (rTMS)
* Conditions that preclude assessing brain function by fMRI: previous head injury, brain surgery, dementia, spinal cord injury, traumatic brain injury, cortical atrophy, serious neurological or medical illness, psychiatric illness, development disability, sensory impairment such as vision and hearing loss, history of birth weight less than 2000 grams and/or gestational age less than 34 weeks)
* MRI compatibility: No major contraindication to MRI (e.g. claustrophobia, pacemaker, vascular stents, metallic ear tubes) and metal implants that would preclude use of MRI
* History of spine surgery with existing instrumentation failure (i.e., broken screws or rods) or pseudarthrosis (lack of fusion) that could be the cause of CLBP
* Any other comorbidity or condition that, in the opinion of the Investigator would make the subject unsuitable for the study or unable to comply with the study requirements

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-04-11 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Detection of brain connectivity using functional MRI | 1 year
  The primary objective of this study is to determine the effects of spinal cord stimulation on chronic low back pain by comparing the functional changes in the central nervous system as measured by fMRI when the spinal cord stimulator is turned on versus when it is turned off.

SECONDARY OUTCOMES:
Detection of brain waves using electroencephalography (EEG) | 1 year
  Characterizing EEG changes in chronic low back pain when the spinal cord stimulator is turned on versus when it is turned off.

OTHER OUTCOMES:
Neurological gait kinematics assessment | 1 year
  Characterizing changes in gait kinematics during a 10-minute walk test in chronic low back pain when the spinal cord stimulator is turned on versus when it is turned off.
Neurophysiological functional assessment using somatosensory evoked potential (SSEP) | 1 year
  Characterizing electrophysiological changes in SSEPs to evaluate the neurotransmission of pain when the spinal cord stimulator is turned on versus when it is turned off.
Neurophysiological functional assessment using pain-related evoked potential (PREP) | 1 year
  Characterizing electrophysiological changes in PREPs to evaluate the neurotransmission of pain when the spinal cord stimulator is turned on versus when it is turned off.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel C Lu, MD, PhD, Principal Investigator — University of California, Los Angeles; Lily Chau, MD, PhD, Study Director — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No